CLINICAL TRIAL: NCT03656666
Title: The AP-GELP Study: A Randomized, Placebo-Controlled Clinical Trial on the Effects of Phosphodiesterase 4-Inhibitor Apremilast in Female Genital Erosive Lichen Planus
Brief Title: The AP-GELP Study: A Clinical Trial on the Effects of Apremilast in Female Genital Erosive Lichen Planus
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: Celgene Corporation (Industry); Amgen (Industry)
Responsible Party: Principal Investigator, Anne Lise Helgesen, Principal Investigator, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AP-GELP
Record Dates: First submitted 2018-08-15; First posted 2018-09-04 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Lichen Planus of Vulva; Female Genital Disease
Keywords: apremilast; genital erosive lichen planus
MeSH Terms: conditions — Genital Diseases, Female | interventions — apremilast

STUDY DESIGN:
Intervention Model Description: Double-blinded, randomized, placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Apremilast (Active Comparator): Week 0-24: 21 patients will receive apremilast oral tablets with initial standard titration of dose day 1-6 followed by standard dose of 30 mg apremilast b.i.d.
  Initial titration:
  Day 1: 10 mg in morning. Day 2: 10 mg in morning and 10 mg in evening. Day 3: 10 mg in morning and 20 mg in evening. Day 4: 20 mg in morning and 20 mg in evening. Day 5: 20 mg in morning and 30 mg in evening. Day 6 and thereafter: 30 mg twice daily.
  Interventions: Drug: Apremilast
- Placebo + Apremilast (Placebo Comparator): Week 0-24: 21 patients will receive matching placebo oral tablets, with initial titration.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Apremilast — Apremilast oral tablets
  Other Names: Otezla
  Arms: Apremilast
Drug: Placebo — Placebo oral tablets
  Other Names: Placebo (for apremilast)
  Arms: Placebo + Apremilast

SUMMARY:
Genital erosive lichen planus (GELP) is a chronic inflammatory disease causing painful genital sores and scarring in women. Treatment options are limited and often unsatisfactory. This trial will study the effects of treatment with apremilast and quality of life and sexual function in women with GELP.

DETAILED DESCRIPTION:
Genital erosive lichen planus (GELP) is a chronic, inflammatory and scarring genital disease. The disease may have a significant impact on daily living, quality of life and sexual function. There is a considerable lack of high-quality evidence on treatment options for GELP and few effective therapeutic facilities available in current clinical practice.

The aims of this study are to investigate clinical and immunohistochemical effects of a new oral anti-inflammatory treatment, apremilast, for women with moderate-to-severe GELP in a double-blinded, randomized, placebo-controlled trial (RCT). Apremilast is an inhibitor of phosphodiesterase 4 (PDE4) with documented effect in several inflammatory skin diseases, but it has not yet been studied in patients with GELP. The drug dose and study design have been chosen based on relevant experience from other studies on apremilast, and is equivalent to the dose used for approved indications (chronic plaque psoriasis and psoriatic arthritis).

The main objective of this trial is to assess the efficacy of apremilast in the treatment of GELP in women.

Secondary objectives include

* Description of immunohistochemical changes in lichen planus lesions
* Assessment of safety of apremilast in the treatment of GELP
* Assessment of quality of life and sexual function

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe GELP at inclusion with the diagnosis based on characteristic clinical and/or histological features. Minimum GELP score 5/30 in vagina and/or vulva (scored separately), of which erythema and pain ≥1 are mandatory
* Informed consent from the patient to the protocol and clinical procedures.

Exclusion Criteria:

* Patients receiving other systemic immune modulating therapy
* Concomitant use of strong CYP3A4 enzyme inducers
* Inadequate birth control, pregnancy and/or breast-feeding
* Depression and suicidal ideation
* Patients with severe renal impairment
* Patients with active tuberculosis, serious infections or cancer
* Unexplained and clinically significant weight loss in underweight patients
* Hypersensitivity to the active substance(s) or to any of the excipients
* Hereditary problems of galactose intolerance, lactase deficiency or glucose-galactose malabsorption
* Participating in another trial that might affect the current study or there should be minimum 90 days between participation in another intervention trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2019-09-24 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean GELP score at week 24 in apremilast-treated patients versus placebo-treated patients | 24 weeks
  The GELP (Genital Erosive Lichen Planus) score is a scoring system for clinical assessment of genital erosive lichen planus (GELP) in women. Area of genital involvement, erythema, striae, number of erosions and pain are registered and scored 0-3 (0 is none) for each parameter. Vulval and vaginal involvement is assessed separately, resulting in a maximum GELP score of 30.

SECONDARY OUTCOMES:
Mean GELP score improvement from week 0 to week 24 in all patients | 24 weeks
  The GELP (Genital Erosive Lichen Planus) score is a scoring system for clinical assessment of genital erosive lichen planus (GELP) in women. Area of genital involvement, erythema, striae, number of erosions and pain are registered and scored 0-3 (0 is none) for each parameter. Vulval and vaginal involvement is assessed separately, resulting in a maximum GELP score of 30.
Weekly use of topical steroid, collected from patient diary | 24 weeks
  Frequency of application is recorded once a week in the patient diary as the number of days being used per week
Weekly VAS pain score, collected from patient diary | 24 weeks
  VAS is recorded once a week in the patient diary using a visual linear scale of 100mm ranging from 0 (no pain) to 10 (worst imaginable pain).
Number of patients with GELP score improvement at week 16 and 24 | 24 weeks
  The GELP (Genital Erosive Lichen Planus) score is a scoring system for clinical assessment of genital erosive lichen planus (GELP) in women. Area of genital involvement, erythema, striae, number of erosions and pain are registered and scored 0-3 (0 is none) for each parameter. Vulval and vaginal involvement is assessed separately, resulting in a maximum GELP score of 30.
Separate GELP score assessments: Area of involvement (in cm²) | 24 weeks
  Range 0-3 (none=0, <3 cm²=1, 3-6 cm²=2, >6 cm²=3). Recorded as part of the GELP score at time points specified in the protocol.
Separate GELP score assessments: Intensity of erythema | 24 weeks
  Range 0-3 (none=0, mild=1, moderate=2, strong=3). Recorded as part of the GELP score at time points specified in the protocol.
Separate GELP score assessments: Number of erosions | 24 weeks
  Range 0-3 (none=0, 1=1, 2-3=2, >3=3). Recorded as part of the GELP score at time points specified in the protocol.
Separate GELP score assessments: Striae | 24 weeks
  Range 0-3 (none=0, minimal=1, moderate=2, extensive=3). Recorded as part of the GELP score at time points specified in the protocol.
Separate GELP score assessments: Pressure-induced pain (VAS) | 24 weeks
  Patient-reported pain is induced by pressuring the involved area with a cotton swab, using a visual linear scale of 100mm ranging from 0 (no pain) to 10 (worst imaginable pain). GELP score range 0-3 (no pain=0, VAS 1-3=1, VAS 4-6=2,VAS 7-10=3). Recorded as part of the GELP score at time points specified in the protocol.
Physician Global Assessment (PGA) | 24 weeks
  5-point disease severity scoring system, assessed by the clinician at time points specified in the protocol (0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe).
Patient Global Assessment (PtGA) | 24 weeks
  5-point disease severity scoring system, assessed by the patient at time points specified in the protocol (0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe).
DLQI score | 24 weeks
  The Dermatology Life Quality Index (DLQI) is a 10-question validated questionnaire. Each question is scored 0-3, with a maximum score of 30. The higher the score, the more quality of life is impaired. The time points for DLQI score are specified in the protocol.
GHQ-28 score | 24 weeks
  GHQ-28 is a 28-item version of the General Health Questionnaire (GHQ) subdivided into somatic symptoms, anxiety/insomnia, social dysfunction and severe depression. Each question is scored 0-1. The higher the score, the more severe the condition.The time points for GHQ-28 score are specified in the protocol.
Sexual function assessments | 24 weeks
  The Female Sexual Distress Scale - Revised (FSDS-R) is a 13-item questionnaire used for sexual function assessment. Each question is scored 0-4. The total score range is 0-52, with higher scores indicating more sexually related distress.

OTHER OUTCOMES:
Description of immune histochemical changes and expression of selected cytokines before and after apremilast therapy, assessed in vulvar or vaginal biopsies | 24 weeks
  Asessment in biopsies at week 0 and 24
Description of extragenital lichen planus at week 0, 16 and 24 | 24 weeks
  Extragenital lichen planes is described and compared at 0,16 and 24 weeks
Evaluation of clinical photos | 24 weeks
  Clinical photos of lichen planus lesions are taken by a medical photographer at week 0 and 24
Adverse events | 24 weeks
  Adverse events are registered at time point described in the protocol

CONTACTS AND LOCATIONS:
Overall Officials: Anne Lise Helgesen, MD PhD, Principal Investigator — Oslo University Hospital HF
Locations (1):
- Oslo University Hospital HF, Oslo, Norway